CLINICAL TRIAL: NCT06360276
Title: Empowering Mind-Body Wellness: Effect of Bundling Seated Exercises and Psychoeducational Rehabilitation Using the Teach-Back Approach on Fatigue and Coping of Women Postmastectomy
Brief Title: Effect of Seated Exercises and Psychoeducational Rehabilitation on Fatigue and Coping of Women Postmastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Assisstant Profesor, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14012021
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Fatigue; Coping Behavior
Keywords: Breast cancer; Exercise Intervention; Psychoeducation; Teach-back; Fatigue; Coping
MeSH Terms: conditions — Fatigue; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seated Exercises (Experimental): Women practiced seated exercises
  Interventions: Behavioral: Seated Exercises
- Psychoeducational Rehabilitation (Experimental): Women received psychological rehabilitation
  Interventions: Behavioral: Psychoeducational Rehabilitation
- Routine Care (Active Comparator): Women received routine health education in the unit
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Seated Exercises — A quasi-experimental research was conducted in the main University Hospital, Alexandria, Egypt. women practiced seated exercises
  Arms: Seated Exercises
Behavioral: Psychoeducational Rehabilitation — Women received Psycho-educational Rehabilitation, including mindfulness breathing, problem-solving training, cognitive re-framing technique, and thought stopping.
  Arms: Psychoeducational Rehabilitation
Behavioral: Routine Care — Women received routine health education in the unit, where nurses provided general instructions about the postoperative activities for women with breast cancer.
  Arms: Routine Care

SUMMARY:
This study aimed to examine the effect of bundling seated exercises and psychoeducational rehabilitation using the teach-back approach on fatigue and coping of women postmastectomy.

Hypotheses for research:

1. Women with BC who receive seated exercises and psychoeducational rehabilitation using the teach-back approach after mastectomy exhibit less fatigue than those who do not.
2. Women with BC who receive seated exercises and psychoeducational rehabilitation using the teach-back approach after mastectomy exhibit improved coping behaviors than those who do not.

A quasi-experimental research was conducted in the main University Hospital, Alexandria, Egypt. A total of 60 women were randomly allocated to one of two groups.; women in the study group practiced seated exercises and psychological rehabilitation interventions, including mindfulness breathing, problem-solving training, cognitive reframing technique, and thought stopping.

DETAILED DESCRIPTION:
A quasi-experimental research was conducted in the main University Hospital, Alexandria, Egypt. A total of 60 women were randomly allocated to one of two groups.; women in the study group practiced seated exercises and psychological rehabilitation interventions.

Researchers prepared a health education unit and designed a booklet about seated exercises and psychological interventions. The developed program was applied to each patients using teach-back method.

Seated Exercises In the sitting position, women were instructed to perform different types of exercises. Researchers demonstrated each exercise and asked women to practice preoperatively to be ready for re-demonstrating them after surgery. Patients were asked to perform the exercise repeatedly until mastering the necessary skills.

Psychological Rehabilitation The participants received training about the implementation of four psychological interventions, namely mindfulness breathing, problem-solving training, cognitive reframing, and thought stopping.

Follow-up Women were instructed to practice each exercise ten times and repeat the whole activity five times per day. Women were followed up for two months to ensure their commitment to the program and provide the needed support.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Adult
* Fully conscious
* Having Breast Cancer
* Planned for mastectomy

Exclusion Criteria:

- Hemodynamically unstable

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Piper Fatigue Scale | one month
  The scale was developed to measure the subjective dimension of fatigue. It include 22 items measuring four elements of subjective fatigue: behavioral/temporal (6 items), sensory (5 items), cognitive/mood (6 items), and affective/emotional meaning (5 items). Participants were asked to rate their level of fatigue on a scale ranging from 0 to 10. The total score ranges from 0 to 220; the higher the score, the higher the fatigue level
Mini-Mental Adjustment to Cancer Scale | one month
  This self-report survey created to gauge the cancer patients' ways to cope. It consists of 29 items rated on a four-point Likert scale ranging from 1 "Does not apply at all to me" to 4 "Totally applies to me"). It includes five subscales under two main categories: maladaptive coping, including helplessness/hopelessness (8 items), and anxious preoccupation (8 items). The higher the score, the higher the maladaptive coping. However, adaptive coping includes fighting spirit (4 items), fatalism (5 items), and cognitive avoidance (4 items) . In this category, high scores means increased the likelihood of adaptive coping skills.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Taha, Professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piper BF, Dibble SL, Dodd MJ, Weiss MC, Slaughter RE, Paul SM. The revised Piper Fatigue Scale: psychometric evaluation in women with breast cancer. Oncol Nurs Forum. 1998 May;25(4):677-84. PMID 9599351
- [Background] Czerw A, Religioni U, Szymanski F, Nieradko-Heluszko A, Mekal D, Hering D, Kowalczuk A, Merks P, Borowska M, Bogdan M, Pajewska M. Normalization of the Mini-MAC (Mental Adjustment to Cancer) Questionnaire among Cancer Patients. Int J Environ Res Public Health. 2021 Nov 29;18(23):12603. doi: 10.3390/ijerph182312603. PMID 34886329
- [Result] Ahmadidarrehsima S, Bidmeshki EA, Rahnama M, Babaei K, Afshari M, Khandani BK. The Effect of Self-Management Education by the Teach-Back Method on Uncertainty of Patients with Breast Cancer: a Quasi-Experimental Study. J Cancer Educ. 2020 Apr;35(2):366-372. doi: 10.1007/s13187-019-1474-5. PMID 30680649
- [Result] Brown JC, Huedo-Medina TB, Pescatello LS, Pescatello SM, Ferrer RA, Johnson BT. Efficacy of exercise interventions in modulating cancer-related fatigue among adult cancer survivors: a meta-analysis. Cancer Epidemiol Biomarkers Prev. 2011 Jan;20(1):123-33. doi: 10.1158/1055-9965.EPI-10-0988. Epub 2010 Nov 4. PMID 21051654
- [Result] Choi S, Choi J. Effects of the teach-back method among cancer patients: a systematic review of the literature. Support Care Cancer. 2021 Dec;29(12):7259-7268. doi: 10.1007/s00520-021-06445-w. Epub 2021 Jul 24. PMID 34302545
- [Result] Cipolletta S, Simonato C, Faccio E. The Effectiveness of Psychoeducational Support Groups for Women With Breast Cancer and Their Caregivers: A Mixed Methods Study. Front Psychol. 2019 Feb 18;10:288. doi: 10.3389/fpsyg.2019.00288. eCollection 2019. PMID 30833920
- [Result] Eisenhut L, Sadeghi-Bahmani D, Gerber M, Saemann A, Staub L, Brand S, Cordier D. Effects of two types of exercise training on psychological well-being, sleep and physical fitness in patients with high-grade glioma (WHO III and IV). J Psychiatr Res. 2022 Jul;151:354-364. doi: 10.1016/j.jpsychires.2022.03.058. Epub 2022 May 3. PMID 35537372
- [Derived] Rashwan ZI, Shaheen SR, Rasoul ASAFA, Kamel NMF, Darweesh HAM. Empowering mind-body wellness: effect of bundling seated exercises and psychoeducational rehabilitation using the teach-back approach on fatigue and coping of women postmastectomy. BMC Womens Health. 2024 Aug 6;24(1):443. doi: 10.1186/s12905-024-03242-5. PMID 39107751